CLINICAL TRIAL: NCT03177343
Title: Pristinamycin in the Treatment of MSSA Bone and Joint Infection
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL17_0384
Record Dates: First submitted 2017-06-02; First posted 2017-06-06 (Actual); Last update posted 2017-06-06 (Actual); Status verified 2017-06

CONDITIONS: Methicillin Susceptible Staphylococcus Aureus (MSSA) Infection; Bone and Joint Infection
Keywords: Pristinamycin; Staphylococcus aureus; Bone and joint infection
MeSH Terms: conditions — Infections; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Staphylococcus aureus represents the leading pathogen implicated in bone and joint infection (BJI), usually requiring prolonged combination antimicrobial therapy, which may be particularly challenging in the case of MDR bacteria and/or for patients with multiple drug intolerance. In the absence of new well-tolerated oral antistaphylococcal drugs, older antibiotics must be considered, such as the pristinamycin.

However, pristinamycin is not currently licensed for treatment of staphylococcal BJI and lack of clinical data prevents it from being considered as a reliable alternative therapeutic option in current guidelines.

The aim of this study is to evaluate pristinamycin (efficacy and tolerance) in the treatment of MSSA bone and joint infection (BJI).

ELIGIBILITY:
* Inclusion Criteria:
* All patients receiving pristinamycin as a part of treatment for an MSSA BJI and followed up between 2001 and 2011 in the infectious diseases department of Hospices Civils de Lyon (HCL)
* Exclusion Criteria:
* Patients with BJI related to diabetic foot or decubitus ulcer

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All patients receiving pristinamycin as a part of treatment for an MSSA BJI and followed up between 2001 and 2011 in the infectious diseases department of HCL
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Efficacy of pristinamycin in MSSA bone and joint infection | 80 weeks
  Outcome of patients having had pristinamycin is described in this part. The follow up of the patients after termination of antimicrobial treatment is almost 80 weeks.
  Treatment failure included: persisting infection under appropriate antimicrobial therapy, relapse after interruption of antimicrobial therapy, septic indication for surgical revision > 5 days after primary surgery, superinfection; and/or death, if related to the BJI or to complication of its management.

SECONDARY OUTCOMES:
Tolerance of pristinamycin in MSSA bone and joint infection | 45 weeks
  The treatment duration could be long (several weeks) as pristinamycin is also used as a long-term suppressive therapy in BJI; thus, we can have 45 weeks of treatment with pristinamycin.
  Pristinamycin-related adverse events (AEs) occurring during follow-up were noted and classified according to the Common Terminology Criteria for Adverse Events (CTCAE; National Cancer Institute, 2003). The accountability of pristinamycin in AE onset was left to the clinician's judgement, with the help of a pharmacovigilance specialist in doubtful cases.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon - Hopital de la Croix Rousse - Centre de reference des infection ostéo-articulaires de Lyon, Lyon, France